CLINICAL TRIAL: NCT01821105
Title: A 2 Phase Comparison of Pre-operative CT AND PET Images in the Intraoperative Detection of Disease to a Hand-held Probe, and to an Intraoperative CT Scan in Patients Undergoing Surgery for Metastatic Colorectal Cancer.
Brief Title: 2 Phase Comparison of Pre-operative CT and PET Images for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Edward Martin, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-0375; NCI-2012-01242 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-09; First posted 2013-03-29 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV A Bladder Cancer; Stage IV A Rectal Cancer; Stage IV B Colon Cancer; Stage IV B Rectal Cancer
Keywords: computed tomography; CT scan; positron emission tomography; PET; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Urinary Bladder Neoplasms; Colorectal Neoplasms | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; Diagnosis, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preoperative PET and CT Scans (Experimental): Patients undergo preoperative whole-body PET scans and CT scans of the abdomen and pelvis. Patients then receive fluoro-deoxyglucose (FDG)IV 60-90 minutes prior to surgery and undergo intraoperative CT scans using a handheld probe and computer navigation system.
  Interventions: Procedure: PET Scan; Procedure: CT Scan; Radiation: fludeoxyglucose F 18; Procedure: computer-aided detection/diagnosis

INTERVENTIONS:
Procedure: PET Scan — All patients will receive whole body PET scans (chest-abdomen-pelvis).
Procedure: CT Scan — All patients will receive CT scans of the abdomen and pelvis with contrast.
Radiation: fludeoxyglucose F 18 — Given IV
  Other Names: 18FDG; FDG
Procedure: computer-aided detection/diagnosis — Undergo computer-aided detection/diagnosis during surgery

SUMMARY:
This pilot phase II studies how well computed tomography (CT) and positron emission tomography (PET) imaging works in detecting disease in patients undergoing surgery for metastatic colorectal cancer. Diagnostic procedures, such as CT and PET scans, done before and during surgery may help find colorectal cancer and help guide surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of rigidly (linearly) registering PET to CT images and applying this fused dataset to guide surgery with an image-guided navigation system and a handheld positron probe in order to facilitate disease detection and improve resection accuracy in advanced stage colorectal cancer.

II. To complete development of software for the nonlinear registration of PET and CT datasets.

OUTLINE:

Patients undergo preoperative whole-body PET scans and CT scans of the abdomen and pelvis. Patients then receive 18 F fludeoxyglucose (FDG) intravenously (IV) 60-90 minutes prior to surgery and undergo intraoperative CT scans using a handheld probe and computer navigation system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed colorectal carcinoma and preoperative PET scan with evidence of hypermetabolic lesions suspicious for cancer will be eligible for this study. In cases of primary cancer, there must be a tissue-confirmed diagnosis. In recurrent cases, patients must have clinical evidence by CT or MRI of disease suitable for resection.
* Patients must be candidates for clinically indicated surgery.
* Patients with recurrent disease may have had prior surgery and/or chemotherapy with no limit to the number of prior therapeutic procedures or chemotherapeutic regimens.
* Patients must have a performance status of 0, 1 or 2 by ECOG(Eastern Cooperative Oncology Group)standards.
* Patients must give written informed consent including consent to have IV line placed for FDG administration.
* Patients must be at least 18 years of age. Children under the age of 18 are excluded from the study due to the rarity of colorectal cancer in children.
* Because radiolabeled agents are known to be teratogenic, women of child-bearing potential and men must agree to use an acceptable form of contraception prior to study entry and for the duration of the study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Organ function requirements: Patients must have organ and marrow function adequate to undergo laparotomy. Specifically:
* Serum creatinine < 2.0 mg/dl
* Serum bilirubin < 2.0 mg/dl
* AST(aspartate aminotransferase,serum glutamate oxaloacetate transaminase, serum glutamate oxaloacetate transaminase,serum glutamate pyruvate transaminase)[SGOT]/ALT[SGPT]<4 times institutional upper limit of normal
* Total WBC(white blood cell)>4,000/mm3 or ANC(absolute neutrophil count)> 1,500/mm3
* Platelets > 100,000/mm3
* Hgb >10g/dl
* Patient must have no clinically significant cardiac disease (New York Heart Association Class III/IV); no serious infection requiring treatment with antibiotics; no other serious ill-ness or illness requiring the use of steroids; no clinically significant pulmonary disease or other illness that would contraindicate or increase the risk of complications at surgery.
* Fasting blood sugar less than 120 mg/dl

Exclusion Criteria:

* Patients with active CNS (central nervous system)tumor involvement are ineligible.
* Any patient who has retained childbearing potential will not be pregnant or lactating and must use adequate contraception to assure avoidance of conception.
* Body size prohibits use of the diagnostic equipment (portable CT scanner).
* Tumor burden is so great (as determined by preoperative PET scanning or intraoperative findings) that further surgery is not advised.
* If lesions are detected with preoperative CT but not with PET scanning (in other words, all patients will have a positive PET scan as part of the inclusion criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Martin, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Sarikaya I, Povoski SP, Al-Saif OH, Kocak E, Bloomston M, Marsh S, Cao Z, Murrey DA, Zhang J, Hall NC, Knopp MV, Martin EW Jr. Combined use of preoperative 18F FDG-PET imaging and intraoperative gamma probe detection for accurate assessment of tumor recurrence in patients with colorectal cancer. World J Surg Oncol. 2007 Jul 16;5:80. doi: 10.1186/1477-7819-5-80. PMID 17634125
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preoperative PET and CT Scans
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Preoperative PET and CT Scans
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 54 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 21
Mean time interval from initial treatment to PET scan [Median (Full Range); unit: months] | 42 [3 to 102]
Mean time interval from PET scan to surgery/GP study [Median (Full Range); unit: days] | 16 [1 to 41]

OUTCOME MEASURES:

1. Primary Outcome: Detection of Position Accuracy With Handheld Probe on Anatomical Location.
Time Frame: up to 12 months
Population: number of tumor lesions detected by the probe
Measure: Number; unit: lesions
Units Other Than Participants: Lesions
Arm/Group | Preoperative PET and CT Scans
Number analyzed (Participants) | 21
Number analyzed (Lesions) | 45
lesions
  true postive | 35
  false positive | 8
  not evaluable | 2

2. Secondary Outcome: All Adverse Events and Complications
Time Frame: up to 12 months
Measure: Number; unit: patients
Arm/Group | Preoperative PET and CT Scans
Number analyzed (Participants) | 21
patients | 0

3. Secondary Outcome: Tumor Detection
Time Frame: At surgery
Measure: Number; unit: lesions detected
Arm/Group | Preoperative PET and CT Scans
Number analyzed (Participants) | 21
lesions detected | 48

ADVERSE EVENTS:
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Arm/Group | Preoperative PET and CT Scans
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes